CLINICAL TRIAL: NCT04070989
Title: Multi-Center, Non-controlled, Prospective Radiostereometric Analysis of the Pinnacle Acetabular Shell
Brief Title: Pinnacle RSA Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to terminate early. Decision was not based on safety or efficacy of the study product.
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSJ_2018_02
Record Dates: First submitted 2019-07-24; First posted 2019-08-28 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis; Degenerative Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Posterior Approach (Experimental): Pinnacle Acetabular Shell (Sector, Gription, no screws), AltrX Polyethylene Liner and Corail Femoral Stem implanted via the posterior approach
  Interventions: Device: THA
- Lateral Approach (Experimental): Pinnacle Acetabular Shell (Sector, Gription, no screws), AltrX Polyethylene Liner and Corail Femoral Stem implanted via the lateral approach
  Interventions: Device: THA
- Anterior Approach (Experimental): Pinnacle Acetabular Shell (Sector, Gription, no screws), AltrX Polyethylene Liner and Corail Femoral Stem implanted via the anterior approach
  Interventions: Device: THA

INTERVENTIONS:
Device: THA — Pinnacle Acetabular Shell (Sector, Gription, no screws), AltrX Polyethylene Liner and Corail Femoral Stem

SUMMARY:
The primary objective is to establish the mean superior cup migration of the Pinnacle Acetabular Shell using model-based RSA over the first two years post-implantation. The primary endpoint is the mean vertical subsidence (Y translation, also known as superior cup migration) at 2 years as measured with RSA. This will be summarized for each surgical approach separately, as well as combined.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals requiring primary THA for a severely painful and/or disabled joint from osteoarthritis, traumatic arthritis, rheumatoid arthritis, or congenital hip dysplasia, AVN of the femoral head or acute traumatic fracture of the femoral head or neck
2. Individuals who are able to speak, read and comprehend the informed patient consent document and willing and able to provide informed patient consent for participation in the study and have authorized the transfer of his/her information to DePuy Synthes
3. Individuals who are willing and able to return for follow-up as specified by the study protocol
4. Individuals who are a minimum age of 21 years at the time of consent
5. Individuals who are willing and able to complete the Subject Hip Outcomes questionnaires as specified by the study protocol

Exclusion Criteria:

1. Individuals have active local or systemic infection
2. Individuals who have loss of musculature, neuromuscular compromise or vascular compromise that would impact rehabilitation following surgery
3. Individuals with poor bone quality, such as osteoporosis, where in the surgeon's opinion, there could be considerable migration of the prosthesis or require additional acetabular cup fixation using screws, or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the implant(s)
4. Individuals with Charcot's or Paget's disease
5. Individuals who, in the judgement of the investigator, would not be a candidate for protocol allowable components to be used for their THA
6. Women that are pregnant or lactating
7. Individuals who have had a contralateral hip that was implanted less than 6 months prior to the time of consent into this study or individuals that expect to have a contralateral hip implanted in the following 6 months at the time of consent into this study
8. Individuals that have amputations in either leg that would impact rehabilitation following surgery
9. Individuals who are bedridden.
10. Individuals that have participated in a clinical investigation with an investigational product (drug or device) in the last three months
11. Individuals currently involved in any personal injury litigation, medical-legal or worker's compensation claims
12. Individuals, in the opinion of the Investigator, who are drug or alcohol abusers or have psychological disorders that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements
13. Individuals diagnosed and taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia
14. Subject has a medical condition with less than 2 years life expectancy
15. Individual has a BMI >45 kg/m2.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Concordia Joint Replacement Group, Concordia Hip and Knee Institute & University of Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre & Dalhousie University, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at https://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of total 100 participants enrolled, 84 participants underwent surgery via either posterior, lateral, or anterior approach. The remaining 16 participants were either withdrawn prior to surgery or the study was terminated prior to surgery and thus they were not included in a surgical approach group.
Period: Overall Study
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach
Started | 40 | 20 | 24
Completed | 29 | 10 | 0
Not Completed | 11 | 10 | 24
Not completed — Death | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 7 | 8 | 23
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Inclusion/Exclusion Criteria not met | 2 | 0 | 1
Not completed — Other | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who received total hip arthroplasty (THA) surgery. Participants were analyzed according to the surgical approach applied during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach | Total
Number analyzed (Participants) | 40 | 20 | 24 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.53 (8.85) | 65.0 (9.39) | 60.5 (12.72) | 65.87 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Analysis Set
  Participants
    Female | 20 | 11 | 9 | 40
    Male | 20 | 9 | 15 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Primary Diagnosis [Count of Participants; unit: Participants] — Population: Safety Analysis Set
  Participants
    Osteoarthritis | 5 | 6 | 23 | 34
    Avascular necrosis | 1 | 0 | 1 | 2
    Degenerative Joint Disease | 34 | 14 | 0 | 48
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: Safety Analysis Set
  kg/m2 | 31.19 (6.73) | 30.36 (6.75) | 30.32 (5.43) | 30.74 (6.33)

OUTCOME MEASURES:

1. Primary Outcome: Mean Superior Cup Migration (Subsidence) at 6 Week and 2 Years
Description: RSA measured mean superior cup migration (subsidence: Y translation in mm) at 6 week and 2 years for each surgical approach separately, as well as combined
Time Frame: At 6 week and 2 years
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Overall Population: Pinnacle Acetabular Shell (Sector, Gription, no screws), AltrX Polyethylene Liner and Corail Femoral Stem implanted via the posterior approach, lateral approach and the anterior approach.
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach | Overall Population
Number analyzed (Participants) | 27 | 15 | 22 | 64
mm
  RSA Measured Subsidence (Y-axis Translation) at 6 weeks: number analyzed (Participants) | 27 | 14 | 21 | 62
  RSA Measured Subsidence (Y-axis Translation) at 6 weeks | -0.001 (0.065) | -0.03 (0.094) | -0.036 (0.133) | -0.02 (0.099)
  RSA Measured Subsidence (Y-axis Translation) at 2yrs: number analyzed (Participants) | 22 | 14 | 0 | 32
  RSA Measured Subsidence (Y-axis Translation) at 2yrs | 0.06 (0.292) | 0.045 (0.501) |  | 0.055 (0.362)

2. Secondary Outcome: RSA Measured Subsidence of the Pinnacle Acetabular Shell at 3 Months, 6 Months and 1 Year
Time Frame: At 3 months, 6 months and 1 year
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach | Overall Population
Number analyzed (Participants) | 27 | 15 | 22 | 64
mm
  RSA measured subsidence of the Pinnacle Acetabular Shell at 3 months f/up: number analyzed (Participants) | 15 | 12 | 15 | 42
  RSA measured subsidence of the Pinnacle Acetabular Shell at 3 months f/up | 0.044 (0.11) | -0.065 (0.103) | -0.062 (0.272) | -0.025 (0.187)
  RSA measured subsidence of the Pinnacle Acetabular Shell at 6 months f/up: number analyzed (Participants) | 26 | 14 | 15 | 55
  RSA measured subsidence of the Pinnacle Acetabular Shell at 6 months f/up | 0.13 (0.314) | 0.047 (0.320) | -0.011 (0.192) | 0.07 (0.289)
  RSA measured subsidence of the Pinnacle Acetabular Shell at 1 year f/up: number analyzed (Participants) | 26 | 12 | 12 | 45
  RSA measured subsidence of the Pinnacle Acetabular Shell at 1 year f/up | 0.065 (0.232) | 0.05 (0.377) | -0.12 (0.287) | 0.032 (0.286)

3. Secondary Outcome: Other RSA Measurements (X-Translations)
Description: Other RSA measurements (X translations in mm) at all time points
Time Frame: At 6 weeks, 3 months, 6 months, 1 year, 2 years
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach | Overall Population
Number analyzed (Participants) | 27 | 15 | 22 | 64
mm
  X-axis translations (mm) at 6 weeks: number analyzed (Participants) | 27 | 14 | 21 | 62
  X-axis translations (mm) at 6 weeks | 0.009 (0.082) | -0.016 (0.214) | 0.049 (0.119) | 0.017 (0.134)
  X-axis translations (mm) at 3 months: number analyzed (Participants) | 15 | 12 | 15 | 42
  X-axis translations (mm) at 3 months | -0.085 (0.229) | -0.042 (0.277) | 0.028 (0.321) | -0.033 (0.276)
  X-axis translations (mm) at 6 months: number analyzed (Participants) | 26 | 14 | 15 | 55
  X-axis translations (mm) at 6 months | -0.001 (0.271) | -0.02 (0.3) | 0.113 (0.402) | 0.025 (0.317)
  X-axis translations (mm) at 1 year: number analyzed (Participants) | 26 | 12 | 7 | 45
  X-axis translations (mm) at 1 year | -0.029 (0.284) | 0.06 (0.283) | 0.146 (0.261) | 0.022 (0.282)
  X-axis translations (mm) at 2 years: number analyzed (Participants) | 22 | 10 | 0 | 32
  X-axis translations (mm) at 2 years | -0.057 (0.372) | -0.026 (0.361) |  | -0.047 (0.363)

4. Secondary Outcome: Other RSA Measurements (Z-Translations)
Description: Other RSA measurements (Z translations in mm) at all time points
Time Frame: At 6 weeks, 3 months, 6 months, 1 year, 2 years
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Overall Population (Per Protocol Analysis): Pinnacle Acetabular Shell (Sector, Gription, no screws), AltrX Polyethylene Liner and Corail Femoral Stem implanted via the posterior approach, lateral approach and the anterior approach.
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach | Overall Population (Per Protocol Analysis)
Number analyzed (Participants) | 27 | 15 | 22 | 64
mm
  Z-axis translations (mm) at 6 weeks: number analyzed (Participants) | 27 | 14 | 21 | 62
  Z-axis translations (mm) at 6 weeks | -0.033 (0.134) | -0.06 (0.15) | -0.033 (0.227) | -0.039 (0.172)
  Z-axis translations (mm) at 3 months: number analyzed (Participants) | 15 | 12 | 15 | 42
  Z-axis translations (mm) at 3 months | -0.087 (0.317) | -0.095 (0.379) | 0.127 (0.409) | -0.013 (0.376)
  Z-axis translations (mm) at 6 months: number analyzed (Participants) | 26 | 14 | 15 | 55
  Z-axis translations (mm) at 6 months | -0.023 (0.303) | -0.199 (0.341) | -0.004 (0.759) | -0.063 (0.476)
  Z-axis translations (mm) at 1 year: number analyzed (Participants) | 26 | 12 | 7 | 45
  Z-axis translations (mm) at 1 year | -0.112 (0.234) | 0.014 (0.41) | -0.095 (0.462) | -0.076 (0.325)
  Z-axis translations (mm) at 2 years: number analyzed (Participants) | 22 | 10 | 0 | 32
  Z-axis translations (mm) at 2 years | -0.207 (0.344) | -0.061 (0.466) |  | -0.161 (0.385)

5. Secondary Outcome: Other RSA Measurements (Rotations)
Description: X, Y, and Z rotations in degrees at all time points
Time Frame: At 6 weeks, 3 months, 6 months, 1 year, 2 years
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Overall Per Protocol Analysis Set: Pinnacle Acetabular Shell (Sector, Gription, no screws), AltrX Polyethylene Liner and Corail Femoral Stem implanted via the posterior approach, lateral approach and the anterior approach.
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach | Overall Per Protocol Analysis Set
Number analyzed (Participants) | 27 | 15 | 22 | 64
Degrees
  X-axis Rotation at 6 Weeks: number analyzed (Participants) | 27 | 14 | 21 | 62
  X-axis Rotation at 6 Weeks | 0.023 (0.368) | -0.175 (0.612) | 0.059 (0.55) | -0.009 (0.495)
  Y-axis Rotation at 6 weeks: number analyzed (Participants) | 27 | 14 | 21 | 62
  Y-axis Rotation at 6 weeks | 0.035 (0.472) | 0.357 (0.588) | -0.033 (0.372) | 0.085 (0.487)
  Z-axis Rotation at 6 weeks: number analyzed (Participants) | 27 | 14 | 21 | 62
  Z-axis Rotation at 6 weeks | 0.045 (0.35) | 0.135 (0.384) | 0.026 (0.377) | 0.059 (0.364)
  X-axis Rotation at 3 months: number analyzed (Participants) | 15 | 12 | 15 | 42
  X-axis Rotation at 3 months | -0.368 (1.046) | -0.021 (1.311) | -0.201 (0.528) | -0.209 (0.974)
  Y-axis Rotation at 3 months: number analyzed (Participants) | 15 | 12 | 15 | 42
  Y-axis Rotation at 3 months | 0.027 (0.966) | 0.053 (1.715) | 0.054 (0.56) | 0.044 (1.102)
  Z-axis Rotation at 3 months: number analyzed (Participants) | 15 | 12 | 15 | 42
  Z-axis Rotation at 3 months | -0.196 (0.475) | -0.231 (0.71) | 0.343 (1.113) | -0.013 (0.841)
  X-axis Rotation at 6 months: number analyzed (Participants) | 26 | 14 | 15 | 55
  X-axis Rotation at 6 months | -0.241 (0.81) | -0.34 (0.811) | 0.481 (3.181) | -0.069 (1.789)
  Y-axis Rotation at 6 months: number analyzed (Participants) | 26 | 14 | 15 | 55
  Y-axis Rotation at 6 months | 0.137 (0.967) | 0.585 (1.043) | -0.254 (1.693) | 0.145 (1.238)
  Z-axis Rotation at 6 months: number analyzed (Participants) | 26 | 14 | 15 | 55
  Z-axis Rotation at 6 months | 0.062 (0.591) | 0.069 (0.575) | 0.549 (1.68) | 0.196 (1.01)
  X-axis Rotation at 1 year: number analyzed (Participants) | 26 | 12 | 7 | 45
  X-axis Rotation at 1 year | -0.024 (0.575) | 0.343 (1.467) | -0.943 (0.773) | -0.069 (0.988)
  Y-axis Rotation at 1 year: number analyzed (Participants) | 26 | 12 | 7 | 45
  Y-axis Rotation at 1 year | 0.043 (0.494) | -0.272 (1.774) | 0.73 (0.738) | 0.066 (1.049)
  Z-axis Rotation at 1 year: number analyzed (Participants) | 26 | 12 | 7 | 45
  Z-axis Rotation at 1 year | 0.067 (0.523) | -0.033 (0.636) | -0.306 (0.774) | -0.018 (0.596)
  X-axis Rotation at 2 years: number analyzed (Participants) | 22 | 10 | 0 | 32
  X-axis Rotation at 2 years | -0.223 (0.703) | 0.26 (1.392) |  | -0.072 (0.974)
  Y-axis Rotation at 2 years: number analyzed (Participants) | 22 | 10 | 0 | 32
  Y-axis Rotation at 2 years | 0.216 (0.801) | -0.156 (1.406) |  | 0.1 (1.019)
  Z-axis Rotation at 2 years: number analyzed (Participants) | 22 | 10 | 0 | 32
  Z-axis Rotation at 2 years | 0.284 (0.714) | -0.001 (0.793) |  | 0.195 (0.739)

6. Secondary Outcome: Linear Head Penetration
Description: Linear head penetration at 1 year and 2 years for each surgical approach separately was reported.
Time Frame: At 1 year and 2 years
Population: Per Protocol Analysis Set. Here 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure while 'n' (number analyzed) signifies participants evaluable for each timepoint. n=0 signifies no participant was available for the analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach
Number analyzed (Participants) | 27 | 12 | 7
mm
  Linear Head Penetration at 1 year f/up | 0.182 (0.107) | 0.211 (0.09) | 0.286 (0.086)
  Linear Head Penetration at 2 years f/up: number analyzed (Participants) | 22 | 10 | 0
  Linear Head Penetration at 2 years f/up | 0.228 (0.101) | 0.321 (0.192) |

7. Secondary Outcome: Patient Reported Outcome Measures (PROMs)- Harris Hip Score
Description: The Harris Hip Score (HHS) has 10 items with four subscales comprising a minimum of 0 points and a maximum of 100 points with higher scores representing better function and outcomes. The four subscales include: pain severity, activities of daily living, absence of deformity and range of motion. Scoring is done according to the following: 90-100 = excellent, 80-89 = good, 70-79 = fair, 60-69 = poor, and below 60 is a failed result.
Time Frame: Pre Operation (-Day90 to Day 0), At 6 weeks, 3 months, 6 months, 1 year and 2 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach
Number analyzed (Participants) | 27 | 15 | 22
Units on a scale
  HHS at Pre-op | 57.6 (15.14) | 49.47 (20.16) | 61.23 (12.61)
  HHS at 6 weeks follow-up: number analyzed (Participants) | 22 | 12 | 21
  HHS at 6 weeks follow-up | 82.14 (11.52) | 76.67 (15.91) | 86.00 (14.07)
  HHS at 3 months follow-up: number analyzed (Participants) | 12 | 9 | 17
  HHS at 3 months follow-up | 90.08 (10.51) | 89.00 (15.58) | 93.18 (6.11)
  HHS at 6 months follow-up: number analyzed (Participants) | 23 | 9 | 17
  HHS at 6 months follow-up | 91.09 (11.22) | 93.89 (9.51) | 96.71 (5.50)
  HHS at 1 year follow-up: number analyzed (Participants) | 27 | 11 | 6
  HHS at 1 year follow-up | 94.93 (7.95) | 96.27 (6.48) | 100 (0)
  HHS at 2 years follow-up: number analyzed (Participants) | 22 | 9 | 0
  HHS at 2 years follow-up | 93.27 (12.55) | 95.44 (7.99) |

8. Primary Outcome: Patient Reported Outcome Measures (PROMs)- HOOS Jr.
Description: Hip Disability and Osteoarthritis Outcome Score, Joint Replacement (HOOS, JR) is a patient reported joint-specific score designed to evaluate outcomes after total hip arthroplasty. It assesses patient pain (2 items), and functions of daily living (4 items). Response to each item is scored from 0 (none) to 4 (extreme). Raw scores are added up and then converted to an interval score (0-100) using an interval table. The final interval score represents a patients total joint disability where 0 corresponds to total joint disability (worse outcome) and 100 is perfect joint health (best outcome).
Time Frame: Pre Operation (-Day90 to Day 0), At 6 weeks, 3 months, 6 months, 1 year and 2 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach
Number analyzed (Participants) | 27 | 15 | 22
Units on a scale
  HOOS Jr. at Pre-op | 52.61 (11.92) | 54.47 (13.99) | 52.88 (16.63)
  HOOS Jr. at 6 weeks follow-up: number analyzed (Participants) | 26 | 13 | 22
  HOOS Jr. at 6 weeks follow-up | 78.99 (11.68) | 80.22 (14.96) | 75.78 (12.22)
  HOOS Jr. at 3 months follow-up: number analyzed (Participants) | 16 | 11 | 18
  HOOS Jr. at 3 months follow-up | 83.17 (14.02) | 88.37 (13.91) | 89.07 (12.62)
  HOOS Jr. at 6 months follow-up: number analyzed (Participants) | 24 | 10 | 18
  HOOS Jr. at 6 months follow-up | 85.7 (14.98) | 90.64 (14.19) | 89.89 (12.00)
  HOOS Jr. at 1 year follow-up: number analyzed (Participants) | 27 | 12 | 6
  HOOS Jr. at 1 year follow-up | 92.71 (11.22) | 91.7 (15.27) | 97.54 (6.02)
  HOOS Jr. at 2 years follow-up: number analyzed (Participants) | 22 | 9 | 0
  HOOS Jr. at 2 years follow-up | 89.76 (15.98) | 94.5 (7.42) |

9. Primary Outcome: Patient Reported Outcome Measures (PROMs)- FJS-12
Description: The Forgotten Joint Score (FJS-12) is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. The Forgotten Joint Score consists of 12 questions with response ranging from 0 (never) to 4 (mostly). All responses are summed and then divided by the number of completed items. This mean value is subsequently multiplied by 25 to obtain a total score range of 0 to 100. Finally, the score is subtracted from 100, to change the direction of the final score in a way that high scores indicate a high degree of "forgetting" the artificial joint, that is, a low degree of awareness.
Time Frame: At 6 weeks, 3 months, 6 months, 1 year and 2 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach
Number analyzed (Participants) | 27 | 13 | 22
Units on a scale
  FJS-12 Score at 6 weeks follow-up | 54.74 (26.14) | 48.14 (29.7) | 55.88 (28.93)
  FJS-12 Score at 3 months follow-up: number analyzed (Participants) | 16 | 11 | 18
  FJS-12 Score at 3 months follow-up | 63.35 (26.5) | 70.27 (31.71) | 69.26 (29.48)
  FJS-12 Score at 6 months follow-up: number analyzed (Participants) | 24 | 10 | 18
  FJS-12 Score at 6 months follow-up | 67.33 (29.78) | 81.88 (18.94) | 82.64 (20.06)
  FJS-12 Score at 1 year follow-up: number analyzed (Participants) | 27 | 12 | 6
  FJS-12 Score at 1 year follow-up | 82.06 (22.58) | 75.87 (27.91) | 91.95 (10.79)
  FJS-12 Score at 2 years follow-up: number analyzed (Participants) | 22 | 9 | 0
  FJS-12 Score at 2 years follow-up | 82.67 (23.72) | 84.72 (11.02) |

ADVERSE EVENTS:
Time Frame: Day 0 up to 2 years
Description: Safety analysis set included all enrolled participants who received THA surgery. Participants were analyzed according to the surgical approach applied during the study.
Arm/Group | Posterior Approach | Lateral Approach | Anterior Approach
All-Cause Mortality (participants affected / at risk) | 1/40 | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 8/40 | 2/20 | 5/24
Other Adverse Events (participants affected / at risk) | 9/40 | 4/20 | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posterior Approach (N=40) | Lateral Approach (N=20) | Anterior Approach (N=24)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posterior Approach (N=40) | Lateral Approach (N=20) | Anterior Approach (N=24)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 2 | 0 | 0
Incision site discharge (Injury, poisoning and procedural complications) | 2 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Stitch abscess (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Early Termination of the study; study was not terminated due to saftey concerns with the product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04070989/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT04070989/SAP_001.pdf